CLINICAL TRIAL: NCT02319577
Title: Randomized, Phase II Study With Gefitinib Plus Vinorelbine Versus Gefitinib Alone in Patients Affected by Non-small Cell Lung Cancer (NSCLC) With Activating Mutations of EGFR
Brief Title: GEfitinib Plus viNOrelbine in Advanced EGFR Mutated NSCLC. GENOA Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Francesco Grossi, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Genoa trial
Record Dates: First submitted 2014-12-09; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; EGFR; vinorelbine; gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gefitinib plus oral vinorelbine (Experimental): Arm A (21-days cycles until progressive disease or unacceptable toxicity):
  Oral vinorelbine 60 mg/mq on days 1,8 Gefitinib 250 mg daily from day 9 to day 21
  Interventions: Drug: oral vinorelbine; Drug: Gefitinib
- Gefitinib alone (Active Comparator): Arm B (21-days cycles until progressive disease or unacceptable toxicity):
  Gefitinib 250 mg daily from day 1 to day 21
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: oral vinorelbine — Anti-neoplastic drug (PO chemotherapeutical agent, vinka alkaloid)
  Other Names: Navelbine
  Arms: Gefitinib plus oral vinorelbine
Drug: Gefitinib — EGFR tyrosine kinase inhibitor
  Other Names: Iressa

SUMMARY:
A sub-population of patients affected by non-small cell lung cancer (NSCLC) with activating mutations of the epidermal growth factor receptor (EGFR) do not gain benefit from treatment with tyrosine-kinase inhibitors (TKIs). The hypothesis of this study is that the addition of chemotherapy with oral vinorelbine to first-line TKI might result in improved outcomes in EGFR-mutated patients.

DETAILED DESCRIPTION:
In spite of the dramatic improvements obtained with EGFR-TKIs in patients affected by NSCLC with activating mutations of EGFR, a fraction of these patients (about 30%) do not respond to EGFR-TKIs or achieve a response of short duration. It has been suggested that these patients may be affected by additional mutations that confer resistance to EGFR-TKIs in spite of the presence of activating mutations of the EGFR gene. Pre-clinical studies show that the addition of chemotherapy to gefitinib may result in increased anti-proliferative activity, and subsequent clinical studies suggest that the synergic activity of gefitinib and chemotherapy can depend from the employed schedules (concurrent versus sequential). Additionally, data from phase I trials of gefitinib plus vinorelbine revealed a high incidence of severe hematological toxicity with concurrent administration, while sequential schedules resulted in a more manageable safety profile.

On the basis of the aforementioned data, we hypothesize that the sequential combination of vinorelbine and gefitinib might result in improved outcomes (in terms of response and survival) in EGFR-mutated NSCLC over gefitinib alone with acceptable tolerability. The availability of an oral formulation of vinorelbine makes it possible to offer the patients an exclusively oral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* At least 18 years old
* Histologically confirmed NSCLC
* Stage IV disease
* Evidence of activating mutations of EGFR
* Measurable disease (assessed by RECIST 1.1)
* No previous chemotherapy or biological therapy for NSCLC
* Previous radiation treatment is allowed, unless all the eligible target lesions have been irradiated, and provided that at least 2 weeks have passed from the end of radiation therapy to the start of the treatment in the study
* Eastern Cooperative Oncology Group (ECOG) performance status : 0-1
* Adequate baseline bone marrow, hepatic and renal function
* In presence of central nervous system metastases, the patient has to be asymptomatic for at least 4 weeks before starting treatment in the study
* Patients who had received neoadjuvant or adjuvant chemotherapy, or concurrent chemo-radiation for non-metastatic, radically treated NSCLC are considered eligible, provided that they had not received vinorelbine as part of such treatment
* Female patients must provide a negative pregnancy test (serum or urine) prior to treatment

Exclusion Criteria:

* Other malignancies within the last 3 years, with exclusion of non-melanoma skin neoplasms and in-situ carcinoma of the cervix
* Grade III-IV New York Heart Association (HYHA) cardiac dysfunction
* Acute myocardial infarction or pulmonary embolism in the last 6 months
* Brain metastases or meningeal carcinomatosis or spinal cord compression, unless controlled and asymptomatic for at least 30 days before starting study treatment
* HIV positivity or AIDS requiring pharmacological treatment
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 6 months | 6 months; tumor assessment is performed every 6 weeks from randomization until progressive disease
  Progression-free survival is defined as the time from randomization until disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) rate at 1 year (1Y-OS), 2 years (2Y-OS), and 3 years (3Y-OS) | Overall survival assessment is performed at every visit from randomization of each patient until his/her death
  Overall survival is defined as the time from randomization to the date of patient date due to any cause or discontinuation of the study. Each OS rate is calculated at the respective end-point (1 year for 1Y-OS, 2 years for 2Y-OS, and 3 years for 3Y-OS).
Response rate (RR) | tumor assessment is performed every 6 weeks from the start of study treatment until progressive disease
  Assessment is performed by response evaluation criteria in solid tumors (RECIST) version 1.1
Safety profile: Safety will be assessed by medical interview, physical examination, and blood collection for complete blood count on days 1 and 8 and biochemistry | assessment of safety profile is performed at every visit (on day 1 and day 8 of each 21-days cycle) from the start of study treatment until three weeks after its interruption due to intolerance or progressive disease
  Evaluation of the safety profile of gefitinib plus oral vinorelbine as compared to the safety profile of gefitinib alone. Safety will be assessed by medical interview, physical examination, and blood collection for complete blood count on days 1 and 8 and biochemistry (sodium, chloride, potassium, calcium, magnesium, phosphorus, glucose, ammonia, creatinine, alkaline phosphatase, aspartate transaminase, alanine transaminase, γ-glutamyl transpeptidase, lactate dehydrogenase, total and fractioned bilirubin, total proteins, albumin) on day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grossi, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genova, Genova, Italy